CLINICAL TRIAL: NCT02481219
Title: COVGIC20482: A Multicenter, Consecutive, Randomized Study to Optimize the Bowel Preparation Regimen for the PillCam COLON 2 Capsule Endoscopy Procedure
Brief Title: Optimization of the Bowel Preparation Regimen for the PillCam® COLON 2 Capsule Endoscopy Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MA-205
Record Dates: First submitted 2015-05-19; First posted 2015-06-25 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2015-06

CONDITIONS: Colorectal Cancer Screening
Keywords: Polyps; Capsule endoscopy; Bowel preparation regimen; Average risk patients for colorectal cancer screening
MeSH Terms: conditions — Polyps | interventions — Sennosides; Metoclopramide; Erythromycin; Bisacodyl; Diatrizoate Meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bowel preparation regimen -Control (Active Comparator): Regimen includes administration of:
  Drug: 4 Senna tablets 2 days before the procedure, Drug: 2-liters of polyethylene glycol (PEG) on the evening before the procedure Drug: 2-liters of PEG on the morning of the procedure, Drug:10mg Metoclopramide or 250 mg Erythromycin Drug: 2 SUPREP oral sulfate solution Drug: 10mg Bisacodyl suppository.
  Interventions: Device: PillCam® COLON 2 procedure-CONTROL; Drug: Senna tablets; Drug: PEG; Drug: Metoclopramide; Drug: Erythromycin; Drug: SUPREP oral sulfate solution; Drug: Bisacodyl
- Bowel preparation regimen-Test (Experimental): Regimen includes administration of:
  Drug: 4 Senna tablets 2 days before the procedure, Drug: 2-liters of PEG on the evening before the procedure Drug: 2-liters of PEG on the morning of the procedure, Drug:10mg Metoclopramide or 250 mg Erythromycin Drug: 2 SUPREP oral sulfate solution with Gastrografin Drug: 10mg Bisacodyl suppository.
  Interventions: Device: PillCam® COLON 2 procedure-CONTROL; Drug: Senna tablets; Drug: PEG; Drug: Metoclopramide; Drug: Erythromycin; Drug: Bisacodyl; Drug: SUPREP oral sulfate solution with Gastrografin

INTERVENTIONS:
Device: PillCam® COLON 2 procedure-CONTROL
Drug: Senna tablets
Drug: PEG
Drug: Metoclopramide
Drug: Erythromycin
Drug: SUPREP oral sulfate solution
  Arms: Bowel preparation regimen -Control
Drug: Bisacodyl
Drug: SUPREP oral sulfate solution with Gastrografin
  Arms: Bowel preparation regimen-Test

SUMMARY:
This study is designed to determine the optimal bowel preparation regimen for PillCam® COLON 2 Capsule Endoscopy System (CCE) procedures in average risk patients.

Patients will be randomized to receive one of two bowel preparation regimens prior to PillCam CCE.

DETAILED DESCRIPTION:
This is a multicenter, prospective, consecutive, randomized study. Average-risk subjects undergoing CCE without optical colonoscopy will be consecutively enrolled and randomized 1:1 to receive one of two bowel preparation regimens prior to PillCam CCE.

Subjects will be enrolled at 5-10 clinical sites in the United States. Subjects who meet the eligibility criteria will be screened for study participation at a baseline visit and will be evaluated on the procedure day or until capsule excretion. A telephone follow-up will be conducted 5 to 9 days post-capsule ingestion to verify capsule excretion, assess patient well-being, and capture any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 50 and 75 years of age.
2. Subject is classified as average risk per the American Gastroenterological Association Guidelines on Colorectal Cancer Screening: Individuals without a personal or family history of colorectal cancer (CRC) or adenomas, inflammatory bowel disease, or high-risk genetic syndromes.
3. Subject is willing and able to participate in the study procedures and to understand and sign the informed consent.

Exclusion Criteria:

1. Subject with history of polyps (including those identified by computed tomography [CT], optical colonoscopy, sigmoidoscopy, etc.).
2. Subject with history of negative colon assessment (including CT, optical colonoscopy, sigmoidoscopy etc.) within 5 years as these subjects would be defined not requiring screening in this time frame.
3. Subject with suspected or diagnosed with hematochezia, melena, iron deficiency with or without anemia, or any other rectal bleeding, including positive fecal occult blood test of any variety.
4. Subject with any condition believed to have an increased risk of capsule retention such as suspected or known bowel obstruction, stricture, or fistula.
5. Subject with dysphagia or any swallowing disorder.
6. Subject with serious medical conditions that would increase the risk associated with capsule or colonoscopy that are so severe that screening would have no benefit.
7. Subject with a cardiac pacemaker or other implanted electromedical device.
8. Subject expected to undergo MRI examination within 7 days after ingestion of the capsule.
9. Subject with clinical evidence of renal disease, including clinically significant laboratory abnormalities of renal function within the past 6 months, or at any time in the past if not tested within the last 6 months, defined as creatinine, blood urea nitrogen (BUN), and/or glomerular filtration rate (GFR) outside of the local laboratory reference range.
10. Subject with known gastrointestinal motility disorders.
11. Subject with allergies or known contraindication to the medications or preparation agents used in the procedure as described in the relevant instructions for use.
12. Subject with comorbidities which, in the opinion of the investigator, will not be appropriate for the study or the subject has an estimated life expectancy of less than 6 months.
13. Subject is considered to be part of a vulnerable population (e.g. prisoners or those without sufficient mental capacity).
14. Subject is pregnant, suspected pregnant, or is actively breast-feeding. Females of child-bearing potential will be required to provide either a urine pregnancy test or serum pregnancy test as part of the participant's standard of care regardless of their participation in the study (except for subjects who are surgically sterile or are post-menopausal for at least two years).
15. Subject has participated in an investigational drug or device research study within 30 days of enrollment that may interfere with the subject's safety or ability to participate in this study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, Dr., Principal Investigator
Locations (6):
- United States (6):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Indiana University Hospital, Indianapolis, Indiana
  - Indianapolis Gastroenterology and Hepatology, Indianapolis, Indiana
  - Dayton Gastroenterology, Dayton, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Franklin Gastroenterology, PLLC, Franklin, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bowel Preparation Regimen -Control: Regimen includes administration of:
  Drug: 4 Senna tablets 2 days before the procedure, Drug: 2-liters of polyethylene glycol (PEG) on the evening before the procedure Drug: 2-liters of PEG on the morning of the procedure, Drug:10mg Metoclopramide or 250 mg Erythromycin Drug: 2 SUPREP oral sulfate solution Drug: 10mg Bisacodyl suppository.
  PillCam® COLON 2 procedure-CONTROL
  Senna tablets
  PEG
  Metoclopramide
  Erythromycin
  SUPREP oral sulfate solution
  Bisacodyl
- Bowel Preparation Regimen-Test: Regimen includes administration of:
  Drug: 4 Senna tablets 2 days before the procedure, Drug: 2-liters of PEG on the evening before the procedure Drug: 2-liters of PEG on the morning of the procedure, Drug:10mg Metoclopramide or 250 mg Erythromycin Drug: 2 SUPREP oral sulfate solution with Gastrografin Drug: 10mg Bisacodyl suppository.
  PillCam® COLON 2 procedure-Test
  Senna tablets
  PEG
  Metoclopramide
  Erythromycin
  Bisacodyl
  SUPREP oral sulfate solution with Gastrografin
Period: Overall Study
Arm/Group | Bowel Preparation Regimen -Control | Bowel Preparation Regimen-Test
Started | 60 | 62
Completed | 58 | 61
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bowel Preparation Regimen -Control: Regimen includes administration of:
  Drug: 4 Senna tablets 2 days before the procedure, Drug: 2-liters of PEG on the evening before the procedure Drug: 2-liters of PEG on the morning of the procedure, Drug:10mg Metoclopramide or 250 mg Erythromycin Drug: 2 SUPREP oral sulfate solution Drug: 10mg Bisacodyl suppository.
  PillCam® COLON 2 procedure-CONTROL
  Senna tablets
  PEG
  Metoclopramide
  Erythromycin
  SUPREP oral sulfate solution
  Bisacodyl
- Total: Total of all reporting groups
Arm/Group | Bowel Preparation Regimen -Control | Bowel Preparation Regimen-Test | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 56 | 114
  >=65 years | 2 | 6 | 8
Age, Continuous [Median (Full Range); unit: years] | 53 [50 to 67] | 53 [50 to 68] | 53 [50 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 29 | 28 | 57
Region of Enrollment [Number; unit: participants]
  United States | 60 | 62 | 122

OUTCOME MEASURES:

1. Primary Outcome: Bowel Cleansing Level of Two Different Bowel Preparation Methods for PillCam® Colon Capsule Endoscopy (CCE)
Description: The primary endpoint is the bowel cleansing level, as determined by a standardized 4-point grading scale, assessed in total and by segment (cecum, ascending, transverse, descending/sigmoid, and rectum).
Time Frame: Within two weeks of study procedure
Population: this was calculated on the per protocol analysis (PPAS) set excluding patients with one (or more) unseen segment in Cecum, Ascending and Transverse colon.
Measure: Number; unit: percentage of particpants
Arm/Group | Bowel Preparation Regimen -Control | Bowel Preparation Regimen-Test
Number analyzed (Participants) | 44 | 54
percentage of particpants
  Overall Excellent cleansing | 6.8 | 16.7
  Cecum Excellent cleansing | 14.0 | 14.6
  Ascending Excellent cleansing | 12.2 | 18.2
  Transverse Excellent cleansing | 10.6 | 14.6
  Descending Excellent cleansing | 9.5 | 18.5
  Rectum Excellent cleansing | 0 | 10.0
  Overall Good cleansing | 70.5 | 59.3
  Cecum Good cleansing | 54.0 | 52.7
  Ascending Good cleansing | 63.3 | 60.0
  Transverse Good cleansing | 61.7 | 60.0
  Descending Good cleansing | 73.8 | 63.0
  Rectum Good cleansing | 56.1 | 52.0
  Overall Fair cleansing | 22.7 | 24.1
  Cecum Fair cleansing | 30.0 | 30.9
  Ascending Fair cleansing | 22.5 | 21.8
  Transverse Fair cleansing | 27.7 | 25.5
  Descending Fair cleansing | 16.7 | 18.5
  Rectum Fair cleansing | 46.5 | 36.0
  Overall Poor cleansing | 0 | 0
  Cecum Poor cleansing | 2.0 | 1.8
  Ascending Poor cleansing | 2.0 | 0
  Transverse Poor cleansing | 0 | 0
  Descending Poor cleansing | 0 | 0
  Rectum Poor cleansing | 2.4 | 2.0

2. Secondary Outcome: Comparing Polyp Detection Rate of Two Different Bowel Preparation Methods for PillCam CCE
Description: Will be assessed from RAPID video in total and by segment
Time Frame: an expected average of 3 weeks from study procedure
Population: This analysis is a subset of the PPAs excluding patients with one or more missing video data for Cecum, Ascending and transverse colon. Patients with at least one polyp detected on overall segments.
Measure: Number; unit: percentage of participants
Arm/Group | Bowel Preparation Regimen -Control | Bowel Preparation Regimen-Test
Number analyzed (Participants) | 47 | 55
percentage of participants
  Overall (any size) | 46.8 | 58.2
  Cecum (any size) | 6.0 | 14.6
  Ascending (any size) | 14.0 | 9.1
  Transverse (any size) | 4.3 | 7.3
  Descending (any size) | 31.9 | 29.1
  rectum (any size) | 24.4 | 32.0
  Overall (polyps ≥6mm) | 21.3 | 36.4
  Cecum (polyps ≥6mm) | 2.0 | 12.7
  Ascending (polyps ≥6mm) | 2.0 | 3.6
  Transverse (polyps ≥6mm) | 4.3 | 7.3
  Descending (polyps ≥6mm) | 12.8 | 16.4
  Rectum (polyps ≥6mm) | 7.3 | 6.0
  Overall (polyps ≥10mm) | 8.5 | 14.6
  Cecum Overall (polyps ≥10mm) | 0 | 7.3
  Ascending Overall (polyps ≥10mm) | 2.0 | 3.6
  Transverse (polyps ≥10mm) | 0 | 1.8
  Descending (polyps ≥10mm) | 4.3 | 3.6
  Rectum (polyps ≥10mm) | 4.9 | 2.0

3. Secondary Outcome: Colonic Transit Time of Two Different Bowel Preparation Methods for PillCam CCE
Description: Colonic transit time of two different bowel preparation was assessed from RAPID video in total and by segment
Time Frame: an expected average of 3 weeks from study procedure
Population: The following patients were excluded from the analysis:2 withdrawn patients, 1 LTF (Lost to follow-up) patient, 2 pattients with failed prcedure, 16 patients with incomplete COLON exam.
Measure: Median (Full Range); unit: hours
Groups:
- Bowel Preparation Regimen - Control: Regimen includes administration of:
  Drug: 4 Senna tablets 2 days before the procedure, Drug: 2-liters of PEG on the evening before the procedure Drug: 2-liters of PEG on the morning of the procedure, Drug:10mg Metoclopramide or 250 mg Erythromycin Drug: 2 SUPREP oral sulfate solution Drug: 10mg Bisacodyl suppository.
  PillCam® COLON 2 procedure-Control
  Senna tablets
  PEG
  Metoclopramide
  Erythromycin
  SUPREP oral sulfate solution
  Bisacodyl
- Bowel Preparation Regimen-Test: Regimen includes administration of:
  Drug: 4 Senna tablets 2 days before the procedure, Drug: 2-liters of PEG on the evening before the procedure Drug: 2-liters of PEG on the morning of the procedure, Drug:10mg Metoclopramide or 250 mg Erythromycin Drug: 2 SUPREP oral sulfate solution with Gastrografin Drug: 10mg Bisacodyl suppository.
  PillCam® COLON 2 procedure- Test
  Senna tablets
  PEG
  Metoclopramide
  Erythromycin
  Bisacodyl
  SUPREP oral sulfate solution with Gastrografin
Arm/Group | Bowel Preparation Regimen - Control | Bowel Preparation Regimen-Test
Number analyzed (Participants) | 46 | 55
hours | 2.8 [0.4 to 7.5] | 2.4 [0 to 5.5]

4. Secondary Outcome: Comparing of Completion Rate of Capsule of Two Different Bowel Preparation Methods for PillCam CCE
Description: Will be assessed from RAPID video in total and by segment
Time Frame: an expected average of 3 weeks from study procedure
Population: Per protocol analysis set
Measure: Number; unit: percentage of participants
Groups:
- Bowel Preparation Regimen -Control: Regimen includes administration of:
  Drug: 4 Senna tablets 2 days before the procedure, Drug: 2-liters of PEG on the evening before the procedure Drug: 2-liters of PEG on the morning of the procedure, Drug:10mg Metoclopramide or 250 mg Erythromycin Drug: 2 SUPREP oral sulfate solution Drug: 10mg Bisacodyl suppository.
  PillCam® COLON 2 procedure- Control
  Senna tablets
  PEG
  Metoclopramide
  Erythromycin
  SUPREP oral sulfate solution
  Bisacodyl
Arm/Group | Bowel Preparation Regimen -Control | Bowel Preparation Regimen-Test
Number analyzed (Participants) | 52 | 55
percentage of participants | 76.9 | 90.9

5. Secondary Outcome: Excretion Rate of Capsule Within 12 Hours of Two Different Bowel Preparation Methods for PillCam CCE
Description: Will be assesses by applicable case report form (CRF)
Time Frame: an expected average of 3 weeks from study procedure
Population: PPAS: Subjects withdrawn prior to the PillCam procedure (3) and subjects with one or more of the following protocol deviations (13) have been excluded: Evening PEG intake <1h and > 2.15h, Morning PEG intake <1h and >2:15 h, Capsule ingestion l<45 min or >75 min after PEG intake , Overall PEG intake volume is less than 3 liters
Measure: Number; unit: percentage of participants
Arm/Group | Bowel Preparation Regimen -Control | Bowel Preparation Regimen-Test
Number analyzed (Participants) | 51 | 55
percentage of participants | 80.4 | 90.9

6. Secondary Outcome: Adverse Events Rate Between Two Different Bowel Preparation Methods for PillCam CCE
Description: Will be assesses by applicable CRF
Time Frame: Adverse Events (AE) were collected starting from the screening visit and until 5-9 days following the PillCam procedure day.
Population: Full analysis set
Measure: Number; unit: percentage of participants with >1 AE
Arm/Group | Bowel Preparation Regimen -Control | Bowel Preparation Regimen-Test
Number analyzed (Participants) | 59 | 62
percentage of participants with >1 AE | 3.4 | 19.4

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected starting from the screening visit and until 5-9 following the PillCam procedure day.
Arm/Group | Bowel Preparation Regimen -Control | Bowel Preparation Regimen-Test
Serious Adverse Events (participants affected / at risk) | 0/59 | 1/62
Other Adverse Events (participants affected / at risk) | 2/59 | 12/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bowel Preparation Regimen -Control (N=59) | Bowel Preparation Regimen-Test (N=62)
Chronic Sinusitis (Eye disorders) | 0 (0) | 1 (1) — Subject experienced double vision and swollen eye and was hospitalized. He was scheduled to undergo Functional Endonasal sinus surgery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bowel Preparation Regimen -Control (N=59) | Bowel Preparation Regimen-Test (N=62)
abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Irritation (General disorders) | 0 (0) | 2 (2) — Skin irritation
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Muscle strain
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)
Haedache (Nervous system disorders) | 1 (1) | 2 (2)
Eye swelling (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior written consent is required for PI to independently publish any study results before a multi-center publication is released. If a multi-center manuscript is not submitted for publication within 1 year after completion of the Trial, PI shall have the right to Publish results. Sponsor shall respond within 45 days and shall have the right to delay the Publication for an additional 90.